CLINICAL TRIAL: NCT05385302
Title: Sociological Determinants of Adherence to Continuous Positive Airway Pressure In the Management of Sleep Apnea Syndrome - A Transdisciplinary Approach.
Brief Title: Sociological Determinants of Positive Airway Pressure Adherence in OSA Patients
Acronym: SOCIO-SAS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: ODENORE (Unknown); HP2 Laboratory (Unknown)
Responsible Party: Sponsor
Other Study IDs: 38RC21.0367
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Adherence, Treatment; Health Literacy; Obstructive Sleep Apnea
Keywords: Adherence; treatment refusal; CPAP; Obstructive sleep apnea; Health literacy
MeSH Terms: conditions — Treatment Adherence and Compliance; Sleep Apnea, Obstructive; Treatment Refusal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicentric, prospective, opened study to evaluate the impact of Health Literacy Levels on CPAP withdrawal in Obstructive Sleep Apnea patients within 6 months of inclusion.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSA) is a chronic multi-organ pathology and heterogeneous in its presentation and phenotypes.

To date, continuous positive airway pressure (CPAP) is the first-line treatment for OSA. In France, 1.2 million patients are treated with CPAP but 15% of patients refused the device at the time of diagnosis and the rate of non-adherence reach 43% 3 years after CPAP initiation.

Both in terms of sleepiness and cardiovascular symptoms, clinical improvement is correlated with normalization of ventilation and therefore with the use of CPAP throughout the sleep period by the patients. Adherence to CPAP is nowadays achieved by the contribution of tele-observance, which provides prescribers, home health care providers and patients with daily feedback on the effectiveness and compliance of the therapy.

To date, studies targeting the predictive factors of CPAP compliance in OSA patients mainly include clinical data (age, sex, severity of OSAS, symptoms, etc.), or technical factors directly related to CPAP treatment (type of mask, residual apnea hypopnea index (AHI) under treatment, leakage, side effects, etc.).

The social, socioeconomic and psychological approaches are far less studied and frankly underestimated, although they are gradually gaining interest, representing the submerged part of the iceberg. Some studies have shown an association between poor socioeconomic status and poor compliance with CPAP, while others have focused on psychological factors. Finally, in the work of our team, we have recently looked at the impact of the marital on compliance and the perception of the associated benefit. However, each study targets a specific area, without taking into account the clinical and individual determinants. Therefore, there is a lack of knowledge about individual determinants of CPAP adherence.

Health literacy, defined as "the ability to access, understand, evaluate, and communicate information in ways that promote, maintain, and improve one's health in a variety of settings across the lifespan" is a possible important limitation for a patient to understand the need for PAP treatment and was never explored in view to explain CPAP adherence.

This project aims to exploit a unique transdisciplinary approach to characterize refusal, discontinuation, and nonadherence to CPAP in patients with diagnosed OSA newly managed on CPAP.

The main hypothesis of the study is that a patient with an insufficient level of health literacy (LS) (score from 0 to 8 defined from the European Health Literacy Survey questionnaire) has a greater probability of stopping treatment early or of being non-compliant than a patient with better performance in terms of health literacy.

ELIGIBILITY:
Inclusion Criteria:

* Patient newly diagnosed with OSA
* Patient with indication for CPAP
* Voluntary patient with informed consent and no objection to participation
* Patient affiliated with or benefiting from a social security plan

Non-Inclusion Criteria:

* Person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure (patient under guardianship or curators) according to articles L1121-5 to L1121-8
* Refusal of participation by the patient
* Patient refusing telemonitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obstructive Sleep Apnea patients with cPAP indication
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
To study the impact of health literacy levels on CPAP discontinuation in newly fitted OSA patients | Between initiation of CPAP (day 7 to 15 after inclusion) to V2 (6 months after inclusion)
  Proportion of CPAP treatment discontinuation without switch to mandibular advancement orthosis treatment

SECONDARY OUTCOMES:
To study the impact of health literacy levels on CPAP refusal after diagnosis. | At V1 (inclusion)
  Proportion of CPAP refusals after diagnosis
To investigate the impact of health literacy levels on adherence status. With adherence status defined here in several ways (≥4h vs <4h; adherence quartiles or adherence clusters). | At 6 month (V2)
  Average CPAP adherence
To study the interactions between the different socio-economic factors studied and their influence on adherence to the CPAP treatment | At 6 month
  Average CPAP adherence
Define the relationship between various clinical, social, economic, environmental determinants and adherence in addition to health literacy. | At 6 months
  Average CPAP adherence
Identify profiles of patients who refuse CPAP or are non- adherent or who have stopped CPAP according to personal determinants | At 6 months
  Adherent, non-adherent, or discontinued status. With adherence status defined here in several ways (≥ 4 hours per night for at least 70% of the nights ; adherence quartiles or adherence clusters).
Determine adherence trajectories as a function of health literacy and specifically study the specific determinants of adherence. | Over 6 months
  Daily CPAP adherence data obtained by telemonitoring
To decipher the links made by people in treatment discontinuation or qualified as non-observant from the medical point of view, between the different factors of non-observance identified. | within 15 days of refusal of CPAP treatment, or within 15 days of discontinuation of treatment during the 6-month follow-up, or within 15 days of visit 2 for both non-adherent and adherent patients at 6 months.
  Criteria identified on the basis of analyses of the corpus carried out from semi-structured interviews concerning knowledge of the pathology, the relationship with the treatment, the relationship with health professionals, and the life trajectory in terms of health care, making it possible to better understand patients' non-adherence.
Understand how people explain these situations based on their life contexts, representations of the disease and treatment, particularly their understanding of the issues involved. | Within 15 days of refusal of treatment for patients refusing CPAP, or within 15 days of discontinuation of treatment for patients who stopped treatment during the 6-month follow-up, or within 15 days of visit 2 for non-adherent patients at 6 month
  Criteria identified on the basis of analyses of the corpus carried out from semi-structured interviews concerning knowledge of the pathology, the relationship with the treatment, the relationship with health professionals, and the life trajectory in terms of health care, making it possible to better understand patients' non-adherence.
Analyze people's perceptions of their health information practices, their relationship with the medical profession and the role of those involved in their pathology to understanding CPAP treatment | Within 15 days of refusal of treatment for patients refusing CPAP, or within 15 days of discontinuation of treatment during the 6-month follow-up, or within 15 days of visit 2 for all patients at 6 month
  Criteria identified on the basis of analyses of the corpus carried out from semi-structured interviews concerning knowledge of the pathology, the relationship with the treatment, the relationship with health professionals, and the life trajectory in terms of health care, making it possible to better understand patients' non-adherence.
Identify the change in adherent patient's relationship to their treatment and the perceived benefits | Within 6 months of the first interview
  Criteria identified on the basis of analyses of the corpus carried out from semi-structured interviews concerning knowledge of the pathology, the relationship with the treatment, the relationship with health professionals, and the life trajectory in terms of health care, making it possible to better understand patients' adherence.
Describe the evolution of non-adherent patient's situation, the health and potential compensation strategies or alternatives that they have implemented to limit the impact of their untreated OSAS | Within 6 months of the first interview for non-adherent patients
  Criteria identified on the basis of analyses of the corpus carried out from semi-structured interviews concerning knowledge of the pathology, the relationship with the treatment, the relationship with health professionals, and the life trajectory in terms of health care, making it possible to better understand patients' non-adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Bailly, PharmD, PhD, Principal Investigator — Sleep and respiratory diseases Lab, CHU Grenoble Alpes
Locations (2):
- France (2):
  - CHUGA, La Tronche
  - Centre du Sommeil de Grenoble, Saint-Martin-d'Hères

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Benjafield AV, Ayas NT, Eastwood PR, Heinzer R, Ip MSM, Morrell MJ, Nunez CM, Patel SR, Penzel T, Pepin JL, Peppard PE, Sinha S, Tufik S, Valentine K, Malhotra A. Estimation of the global prevalence and burden of obstructive sleep apnoea: a literature-based analysis. Lancet Respir Med. 2019 Aug;7(8):687-698. doi: 10.1016/S2213-2600(19)30198-5. Epub 2019 Jul 9. PMID 31300334
- [Derived] Bailly S, Foote A, Mendelson M, Rakotovao A, Borel JC, Pepin JL, Tamisier R, Revil H. Sociological determinants of adherence to continuous positive airway pressure in the management of sleep apnoea syndrome: protocol for a transdisciplinary, prospective observational study. BMJ Open. 2024 Mar 5;14(3):e079765. doi: 10.1136/bmjopen-2023-079765. PMID 38448064